CLINICAL TRIAL: NCT02098642
Title: Passive Mobilization of the Metatarsophalangeal Joint of the Hallux During a Rehabilitation Treatment in Patients With Parkinson's Disease
Brief Title: Hallux Mobilization in Patients With Parkinson's Disease
Acronym: HalluxPD001
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: HalluxPD001; Hallux PD 001 (Other: Ospedale Generale di Zona "Moriggia-Pelascini")
Record Dates: First submitted 2014-03-21; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
Keywords: Gait Disturbances; Metatarsophalangeal joint
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with passive joint mobilization: Patients diagnosed with PD according to the Gelb et al in Hoen&Yahr stage 3, with Freezing of Gait and treated with a Multidisciplinary intensive rehabilitation treatment (MIRT), including the mobilization of the metatarsophalangeal joint of the hallux
  Interventions: Other: MIRT; Other: Mobilization of the metatarsophalangeal joint of the hallux
- No passive joint mobilization: Patients diagnosed with PD according to the Gelb et al in Hoen&Yahr stage 3, with Freezing of Gait and treated with a Multidisciplinary intensive rehabilitation treatment (MIRT)
  Interventions: Other: MIRT

INTERVENTIONS:
Other: MIRT — A 4-week cycle of physiotherapy that entailed three daily sessions, 5 days a week. The first session comprised cardiovascular warm-up activities, relaxation exercises, muscle-stretching, exercises to improve the range of motion of spinal, pelvic and scapular joints, and exercises to improve the functionality of abdominal muscles and postural changes in the supine position. The second session included exercises to improve balance and gait using a stabilometric platform with a visual cue and treadmill training associated with auditory and visual cues (treadmill plus). The last was an occupational therapy session with the aim of improving autonomy in daily living activities.
Other: Mobilization of the metatarsophalangeal joint of the hallux — MIRT and mobilization of the metatarsophalangeal joint of the hallux
  Groups: Patients with passive joint mobilization

SUMMARY:
Parkinson's disease is a degenerative disorder of the central nervous system. The motor symptoms of Parkinson's disease result from the death of dopamine-generating cells in the substantia nigra, a region of the midbrain; the cause of this cell death is unknown. Early in the course of the disease, the most obvious symptoms are movement-related; these include shaking, rigidity, slowness of movement and difficulty with walking and gait. A multidisciplinary intensive rehabilitation treatment (MIRT) is able to improve different parameters in PD that are poorly responsive to dopaminergic therapy. In this study, we aim to understand whether the passive mobilization of the metatarsophalangeal joint of the hallux determines an increase in the joint range in this district, allowing to improve, at least, the gait.

DETAILED DESCRIPTION:
Parkinson's disease is a degenerative disorder of the central nervous system. The motor symptoms of Parkinson's disease result from the death of dopamine-generating cells in the substantia nigra, a region of the midbrain; the cause of this cell death is unknown. Early in the course of the disease, the most obvious symptoms are movement-related; these include shaking, rigidity, slowness of movement and difficulty with walking and gait. The main families of drugs useful for treating motor symptoms are levodopa dopamine agonists and Monoamine oxidases-B inhibitors.A multidisciplinary intensive rehabilitation treatment (MIRT) is able to improve different parameters in PD that are poorly responsive to the pharmacological therapy. In this study, we aim to understand whether the passive mobilization of the metatarsophalangeal joint of the hallux determines an increase in the joint range in this district, allowing to improve, at least, the gait in patients with PD. In this course, we will evaluate whether passive mobilization of this joint, lead to positive effects on the freezing of gait and on the festination.

ELIGIBILITY:
Inclusion Criteria:

PD patients stage 3 H&Y with FOG

Exclusion Criteria:

we excluded patients with atypical parkinsonism, with other concomitant neurological conditions (with cerebrovascular etc.), with joint disorders, muscle disorders or with other orthopedic conditions.

Ages: 49 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
FOGQ | One month
  Freezing of Gait Questionnaire Value

SECONDARY OUTCOMES:
UPDRS III | One month
  Unified Parkinson's disease Rating Scale
BBS | One month
  Berg Balance Scale
Hallux | One month
  Range of metatarsophalangeal joint value

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale Generale Di Zona Moriggia-Pelascini
Locations (1):
- Parkinson's Disease and Movement Disorders Rehabilitation Unit, Gravedona, Como, Italy